CLINICAL TRIAL: NCT07100613
Title: Efficacy of a Microparticulate Muco-adhesive Patch Containing Drug-nutraceutical Association in paTIents Affected by Oral Mucosa Alterations (EMPATIA)
Brief Title: Mucoadhesive Modified-Release Formulations for the Topical Treatment of Symptomatic Oral Lichen Planus
Acronym: EMPATIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Vera Panzarella, Associate Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMPATIA
Record Dates: First submitted 2025-07-19; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Oral Lichen Planus; Oral Lichen Planus Related Stress; Oral Mucosal Disease; Oral Pain
Keywords: mucoadhesive patch; oral lichen planus; clobetasol; resveratrol; drug delivery system; Optical coherence tomography; Ora pain
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Clobetasol; Resveratrol; Orabase

STUDY DESIGN:
Intervention Model Description: Model Description:
  Triple-arm, parallel assignment model with 1:1:1 randomization. Each participant is randomly assigned to one of three intervention groups receiving either: (1) a mucoadhesive patch with clobetasol, (2) a mucoadhesive patch with clobetasol and resveratrol, or (3) clobetasol 0.05% in an orabase-type paste.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clobetasol Patch (Experimental): Participants will receive a mucoadhesive patch containing clobetasol propionate 0.05%. The patch is applied directly to the symptomatic oral lesion once daily for 30 days, following oral hygiene. No food or drink is allowed for 30 minutes after application. The patch is self-dissolving.
  Interventions: Drug: Clobetasol Patch
- Clobetasol + Resveratrol Patch (Experimental): Participants will receive a mucoadhesive patch containing clobetasol propionate 0.05% and resveratrol. The patch is applied once daily for 30 days on the symptomatic oral lesion. It is self-adhering and dissolves without removal. No food or drink is allowed for 30 minutes after application.
  Interventions: Drug: Clobetasol + Resveratrol Patch
- Clobetasol in Orabase (Active Comparator): Participants will receive clobetasol propionate 0.05% in an orabase-type adhesive paste, applied once daily for 30 days after oral hygiene. Application is made directly to the lesion. No food or drink is allowed for 30 minutes after application.
  Interventions: Drug: Clobetasol in Orabase

INTERVENTIONS:
Drug: Clobetasol Patch — A mucoadhesive patch containing clobetasol propionate 0.05%. Applied once daily for 30 days to the oral lesion.
  Other Names: Mucoadhesive Clobetasol Patch
  Arms: Clobetasol Patch
Drug: Clobetasol + Resveratrol Patch — A mucoadhesive patch containing clobetasol propionate 0.05% and resveratrol. Applied once daily for 30 days to the oral lesion.
  Other Names: Mucoadhesive Patch with Clobetasol and Resveratrol
  Arms: Clobetasol + Resveratrol Patch
Drug: Clobetasol in Orabase — Clobetasol propionate 0.05% in orabase-type adhesive paste. Applied once daily for 30 days to the oral lesion.
  Other Names: Clobetasol 0.05% Orabase Paste
  Arms: Clobetasol in Orabase

SUMMARY:
The goal of this clinical trial is to learn if a mucoadhesive patch containing clobetasol alone or in combination with resveratrol can reduce symptoms and improve quality of life in adults with Oral Lichen Planus (OLP). The main questions it aims to answer are:

Does the patch reduce oral pain and burning sensations? Does it improve the appearance of oral lesions and patients' daily well-being?

Researchers will compare:

A patch containing clobetasol A patch containing clobetasol and resveratrol A standard clobetasol 0.05% ointment in an adhesive base

Participants will:

Apply their assigned treatment to the oral lesion daily for 30 days Attend three clinical visits for evaluations and imaging Complete questionnaires about pain, symptoms, and treatment experience

DETAILED DESCRIPTION:
Oral Lichen Planus (OLP) is a chronic inflammatory condition affecting the oral mucosa, often causing painful lesions, burning sensations, and impaired quality of life. Current treatments primarily rely on high-potency topical corticosteroids, such as clobetasol propionate. However, conventional formulations like ointments or pastes may be difficult to apply, poorly retained in the oral cavity, and associated with limited bioavailability or side effects.

This clinical trial investigates the efficacy of a novel mucoadhesive drug delivery system in the form of a patch. The patch is designed to adhere to the oral mucosa, releasing the active compounds in a controlled and prolonged manner. Two types of patches are tested: one containing clobetasol propionate alone and one containing a combination of clobetasol and resveratrol, a natural polyphenol known for its anti-inflammatory and immunomodulatory properties.

The study is a triple-blind, randomized, controlled clinical trial conducted on adult patients with a confirmed histological diagnosis of symptomatic OLP. Participants are randomly assigned to one of three arms:

Arm 1: Patch with clobetasol propionate Arm 2: Patch with clobetasol propionate and resveratrol Arm 3 (Control): Clobetasol 0.05% in an orabase-type adhesive paste Treatments are applied over a 30-day period following a standardized schedule. Clinical evaluations take place at baseline, 15 days, and 30 days, and include photographic documentation, symptom scoring with the Visual Analog Scale (VAS), and clinical severity assessment using the Thongprasom score. In addition, participants complete the Oral Health Impact Profile-14 (OHIP-14) questionnaire to evaluate changes in oral-health-related quality of life.

Structural changes in the mucosa are monitored using Optical Coherence Tomography (OCT), a non-invasive imaging technique that allows real-time visualization of tissue layers, providing objective information on epithelial healing and inflammation.

The primary outcomes are reduction in pain and burning symptoms, improvement of lesion severity, and increased quality of life. Secondary outcomes include patient compliance and OCT-based structural improvement. This study aims to offer a more effective, better tolerated, and innovative therapeutic approach for managing oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Clinical suspicion of Oral Lichen Planus (OLP).
* Histological confirmation of OLP based on World Health Organization (WHO) criteria (presence of hyperkeratosis, acanthosis, basal cell degeneration, and a band-like lymphocytic infiltrate in the lamina propria).
* Absence of epithelial dysplasia.
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Previous diagnosis or treatment for OLP.
* Use of topical or systemic corticosteroids in the last 4 weeks.
* Use of medications known to cause lichenoid reactions.
* History of allergic reactions to dental materials (e.g., amalgam).
* Hematological disorders or immunodeficiencies.
* Pregnancy or breastfeeding.
* Current use of immunosuppressive therapies.
* Inability or unwillingness to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom Intensity (Pain/Burning) | Baseline and Day 30
  Patient-reported pain and burning intensity will be measured using the 10-point Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse symptoms.
Change in Clinical Severity of Lesions | Baseline and Day 30
  Clinical improvement will be assessed using the Thongprasom clinical scoring system (score range 0-5, where 0 = no lesion and 5 = severe erosive lesion). Higher scores indicate worse lesion severity. The outcome will measure the change from baseline to day 30.

SECONDARY OUTCOMES:
Change in Oral Health-Related Quality of Life | Baseline and Day 30
  Evaluated using the Oral Health Impact Profile-14 (OHIP-14) questionnaire (range 0-56, with higher scores indicating worse quality of life).
Compliance with Treatment | Day 15 and Day 30
  Adherence to the patch protocol, measured as the number of daily applications recorded in participant diaries.
Epithelial Structural Improvement (OCT Imaging) | Baseline and Day 30
  Changes in mucosal architecture will be assessed using Optical Coherence Tomography (OCT). Improvement is defined as reduction in epithelial discontinuities and inflammatory patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy, Italy